CLINICAL TRIAL: NCT03158428
Title: CSD170202: A Crossover Study to Evaluate the Exposure to Tobacco Constituents From Two Moist Snuff Products
Brief Title: CSD170202: A Study to Evaluate the Exposure to Tobacco Constituents From Two Moist Snuff Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: Inflamax Research Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD170202
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSD170202AA, CSD170202AB Use Group (Experimental): Use of product CSD170202AA exclusively for approximately one week (seven days +1/-2 day) prior to a test visit, followed by use of product CSD170202AB exclusively for approximately one week (seven days +1/-2 day) prior to a test visit.
  Interventions: Other: CSD170202AA; Other: CSD170202AB
- CSD170202AB, CSD170202AA Use Group (Experimental): Use of product CSD170202AB exclusively for approximately one week (seven days +1/-2 day) prior to a test visit, followed by use of product CSD170202AA exclusively for approximately one week (seven days +1/-2 day) prior to a test visit.
  Interventions: Other: CSD170202AA; Other: CSD170202AB

INTERVENTIONS:
Other: CSD170202AA — A moist snuff product
Other: CSD170202AB — A moist snuff product

SUMMARY:
This study will evaluate exposure to tobacco constituents from two moist snuff products, and provide a basis for comparing mouth-level exposure (MLE) in moist snuff users after use of each of the two moist snuff products.

DETAILED DESCRIPTION:
This will be an unblinded, single-center, randomized, two-way crossover study, conducted in generally healthy, adult moist snuff users who will be randomly assigned to the order in which they will use two moist snuff study products (comparator product, test product). Enrolled subjects will use one of each of the study products exclusively for approximately one week (seven days +1/-2 day) prior to a test visit, with a different product used each week over a two-week period. During each test visit, subjects will use study product ad libitum during a 6-hour period. Expectoration will be collected from the subjects during each product use. The used study product will be collected after use. Blood samples will be collected at each test visit, prior to study product use, for determination of plasma cotinine levels.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) written in English;
2. Generally healthy males and females, 21 years of age or older, at Screening-Enrollment Visit;
3. Self-reports currently using at least two cans of moist snuff per week;
4. Self-reports that moist snuff is the only tobacco- or nicotine-containing product used within 30 days of the Screening-Enrollment Visit;
5. Usual brand (UB) of moist snuff is one of the products specified in the protocol;
6. Used their UB product for ≥ 3 months;
7. Subject is not delaying a decision to quit using moist snuff to participate in the study;
8. Agrees to exclusively use the study products and not use any other tobacco- or nicotine-containing products during the course of the study;
9. Able to safely perform the required study procedures, as determined by the Investigator.

Exclusion Criteria:

1. Self-reported history of heart disease, kidney disease, diabetes, liver disease, uncontrolled hypertension, or uncontrolled hypercholesterolemia;
2. At risk for heart disease, i.e., obesity (body mass index [BMI] > 43 kg/m2), as determined by the Investigator;
3. Females ≥ 35 years of age currently using systemic, estrogen-containing contraception, or hormone replacement therapy;
4. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to the Screening-Enrollment Visit;
5. Females who are pregnant or breastfeeding, or plan to become pregnant during the course of the study;
6. Participation in another clinical study within 30 days prior to the Screening-Enrollment Visit. (The 30-day window for each subject will be derived from the date of the last study event in the previous study to the Screening-Enrollment Visit of the current study);
7. Determined by the Investigator to be ineligible for the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Mouth-Level Exposure (MLE) of nicotine per gram (or product) | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Segall, MD, Principal Investigator — Clinical Research Atlanta
Locations (1):
- Clinical Research Atlanta, Stockbridge, Georgia, United States

IPD SHARING:
Plan to Share IPD: No